CLINICAL TRIAL: NCT04280250
Title: Can Implementation Intentions Help People Who Are Supported by Secondary and Tertiary Care Mental Health Services to be Less Sedentary and More Physically Active: A Feasibility and Acceptability Study.
Brief Title: Can an Action-based Help-sheet Help People to Move More and Sit Less.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Stephanie Roebuck, Trainee Clinical Psychologist, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NHS00164
Record Dates: First submitted 2020-01-31; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Sedentary Behavior
Keywords: Implementation Intention; If-Then plan; Tertiary mental health services; Secondary mental health services
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Active control arm: Volitional help-sheet with instruction: We want you to plan to increase your level of physical activity. Research shows that if people can identify situations in which they are likely to be tempted not to be physically active and ways to overcome temptation they are much more likely to be successful in their intention to increase their level of physical activity. On the left hand side of the page are a series of common situations in which people feel tempted not to be physically active; please tick all those that apply to you personally. On the right hand side of the page are a series of possible solutions; please tick all those that apply to you personally. Tick as many or as few situations and solutions as you like.
  Interventions: Other: Control condition
- Group 2 (Experimental): Experimental arm: Volitional help-sheet with instruction:
  We want you to plan to increase your level of physical activity. Research shows that if people link being tempted not to be physically active with a way to overcome that temptation, they are much more likely to be successful in their intention to increase their level of physical activity. On the left hand side of the page below is the temptation not to be physically active; on the right hand side of the page are a series of possible solutions. Please draw lines linking being tempted not to be physically active (left hand side) to solutions (right hand side) that you think might work for you personally. Please make as many situation-solution links as you like.
  Interventions: Other: Volitional Help-Sheet

INTERVENTIONS:
Other: Volitional Help-Sheet — Self-help sheet in order to form implementation intentions
  Arms: Group 2
Other: Control condition — Psychoeducational self-help sheet
  Arms: Group 1

SUMMARY:
Implementation intentions support people to turn intentions into action, and "Volitional Help-Sheets" are a tool which helps people to form implementation intentions. The study will recruit participants from secondary and tertiary mental health services. The participants will be randomised to one of two groups. Participants in Group 1, the control group, will receive the Volitional Help-Sheet (psychoeducational self-help sheet) but not form implementation intentions. Participants in Group 2, the experimental condition, will use the Volitional Help-Sheet to form implementation intentions. Participants will then complete an acceptability and feasibility measure. At follow up, participants will repeat baseline measures. The feasibility and acceptability of using a Volitional Help-Sheet to form implementation intentions to help people using secondary and tertiary care mental health services to reduce sedentary behaviour will be evaluated.

DETAILED DESCRIPTION:
Introduction: Sedentary behaviour is risk factor for developing many health conditions. People with mental health difficulties can be more sedentary and live 10 years fewer than other populations. Implementation intentions support people to turn intentions into action, and Volitional Help-Sheets are a tool which helps people to form implementation intentions, by identifying critical situations and linking these to potential solutions. The feasibility and acceptability of using a Volitional Help-Sheet to help people using secondary and tertiary care mental health services to reduce sedentary behaviour will be evaluated. If Volitional Help-Sheets are feasible and acceptable to use in this population, this will justify further research in this area, as improving physical and psychological health could increase life expectancy.

Design: The study includes two timepoints: baseline and follow up (four weeks post baseline). Participant characteristics/demographics collected at baseline. At both baseline and follow up, all participants will be asked to complete measures of sedentary behaviour, physical activity, well-being, motivation and mental health. Participants will be randomised to one of two groups. Participants in Group 1, the control group, will receive the Volitional Help-Sheet as a psychoeducational self-help sheet, but not form implementation intentions. Participants in Group 2, the experimental condition, will use the Volitional Help-Sheet to form implementation intentions. Participants will then complete an acceptability and feasibility measure. At follow up, participants will repeat baseline measures.

Sample size: Participants will be current service users, recruited from NHS based secondary and tertiary care mental health services. The recruitment of a minimum of 24 participants and a maximum of 32 participants would be considered a feasible two-armed study.

Recruitment: Adults: 18years+, motivated to decrease sedentary behaviour (demonstrated by choosing to make contact with the researcher to indicate an interest in participation in the study), has capacity to consent to study, currently receiving support from any secondary or tertiary care mental health service and English language ability sufficient to be able to meet the requirements of the study.

Procedure: Recruitment posters will be displayed in clinical areas as part of recruitment. Care teams can advise interested participants on how to contact the researcher and support this if required. Participant information sheets will be disseminated to interested parties. Where a service user has informed the researcher of their interest in participating in the study, they will be offered a detailed participant information sheet and consent to contact forms outlining the study, the expected benefits and commitment required, and informed consent forms. Interested participants will be assessed for capacity to consent and eligibility and will begin the randomisation procedure upon booking the baseline assessment appointment. All members of the research team have experience of obtaining informed consent in research and clinical roles.

Participants will be block randomised (sampling without replacement) in blocks of four and stratified according to clinical service using an online program, into either a control group (group 1) or an experimental arm (group 2). Participants in Group 1 (control arm) will receive a Volitional Help-Sheet with an instruction to tick all situations in which they are tempted not to be active, and tick all solutions to overcome these. Participants in Group 2 (experimental arm) will use the Volitional Help-Sheet to form implementation intentions by linking situations in which they are tempted not to be physically active, with solutions to overcome these. Researchers will be unblinded, however the participants and those external to the research team where involved will remain blind to the group allocated.

Outcomes and analysis: The main study hypothesis is that forming implementation intentions using the Volitional Help-Sheet will be considered acceptable to the participants involved in the study, and that forming implementation intentions using the Volitional Help-Sheet will be considered feasible to use within a diverse range of NHS settings. An exploratory hypothesis is also that the increase in activity will be significantly greater in the treatment group than the control group. Quantitative analysis will be used to evaluate the feasibility and acceptability of using a Volitional Help-Sheet to help people using secondary and tertiary care mental health services to form implementation intentions, with the aim of a reduction in sedentary behaviour.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Motivated to decrease sedentary behaviour (demonstrated by choosing to make contact with the researcher to indicate an interest in participation in the study
* Has capacity to consent to study
* Currently receiving support from any secondary or tertiary care mental health service
* English language ability sufficient to be able to meet the requirements of the study

Participants will not be recruited on the basis of an assumption that they are sedentary, and participants must demonstrate a desire to increase their sedentary behaviour as indicated by choosing to make contact with the researcher to indicate an interest in participation in the study.

Exclusion Criteria:

* Cannot give informed consent
* English language not sufficient to be able to meet the requirements of the study
* Does not meet other criteria for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM). (Weiner et al, 2017) | Change from Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported acceptability measure
Feasibility of Intervention Measure (FIM). (Weiner et al, 2017) | Change from Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported feasibility measure
Intervention Appropriateness Measure (IAM). (Weiner et al, 2017) | Change from Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported appropriateness measure

SECONDARY OUTCOMES:
International Physical Activity Questionnaire short form (Booth, 2000) | Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported physical activity measure
Sedentary Behaviour Questionnaire (Gardener et al, 2011) | Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported sedentary behaviour measure
CORE-OM (Evans et al, 2000) | Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported symptom measure
Office for National Statistics' Measure of Subjective Wellbeing (Dolan, Layard, and Metcalfe, 2011). | Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported wellbeing measure
COM-B measures (Keyworth, Epton, Goldthorpe, Calam, and Armitage, 2019) | Time point 1 (baseline) and Time point 2 (follow up, 4 weeks after baseline)
  Self reported motivation measure

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Roebuck, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.